CLINICAL TRIAL: NCT05893498
Title: Advancing Cath Lab Results With FFRangio Coronary Physiology Assessment
Acronym: ALL-RISE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CathWorks Ltd. (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CathWorks CWX-08
Record Dates: First submitted 2023-04-25; First posted 2023-06-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous Coronary Intervention
Keywords: PCI; Coronary Artery Disease; FFRangio; Pressure Wire-Guided
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FFRangio (Experimental): FFRangio guided revascularization
  Interventions: Device: FFRangio
- Pressure wire (Active Comparator): Pressure wire-based guided revascularization (FFR or NHPR)
  Interventions: Device: FFR or NHPR

INTERVENTIONS:
Device: FFRangio — A 3D image-base software device (CathWorks, Ltd, Kfar Saba, Israel) using three (3) angiographic views to provide a quantitative analysis of the functional significance of coronary lesions.
  Arms: FFRangio
Device: FFR or NHPR — Using an invasive pressure-wire to assess functional significance of coronary lesions either under hyperemic conditions (FFR) or utilizing Non-hyperemic pressure ratios (NHPR).
  Other Names: FFR, iFR RFR, dPR, Pd/Pa
  Arms: Pressure wire

SUMMARY:
To test whether FFRangio-guided treatment is non-inferior to conventional pressure wire-guided treatment in patients with coronary artery disease.

DETAILED DESCRIPTION:
ALL-RISE is a prospective, randomized, multi-center, controlled post-market study. The ALL-RISE study is designed to test whether FFRangio-guided treatment is non-inferior to conventional pressure wire-guided treatment in patients with coronary artery disease being evaluated for percutaneous coronary intervention (PCI) with respect to major adverse cardiac events (MACE) at one year.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ( ≥18 years old) presenting with CCS or NSTEACS with one or more study lesion(s) deemed appropriate (diameter stenosis 50-90%) for both pressure-wire and FFRangio physiologic assessment.

General Exclusion Criteria:

1. Subject with ST-elevation (MI (STEMI) within 72 hours at time of study enrollment
2. Prior coronary artery bypass graft (CABG) with patent grafts to the study vessel(s)
3. Patients undergoing coronary physiologic assessment where one possible outcome is referral for CABG
4. The study vessel supplies a significant nonviable territory (e.g., prior transmural MI)
5. Severe left sided valvular heart disease
6. Most recent documented LVEF ≤30%
7. Women who are pregnant or breastfeeding (women of childbearing potential are required to have negative pregnancy test within 1 week of index procedure)
8. Patients with life expectancy <1 year life as estimated by treating physician.
9. Subjects enrolled in other ongoing non-registry clinical studies that would impact conduct or outcomes of this study (registries and long-term follow-up of other studies are allowed)
10. Subjects who have undergone angiographic or wire-based coronary physiological assessment for 1 or more potential study lesions within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1924 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 1 year
  Rate of the composite of all-cause death, myocardial infarction (MI) or unplanned clinically-driven revascularization

SECONDARY OUTCOMES:
All-Cause Mortality | 12 months
  Total rate of death from any cause
Myocardial Infarction | 12 months
  Total rate of myocardial infarction
Unplanned Revascularization | 12 months
  Total rate of unplanned clinically-driven revascularization
Stent thrombosis | 12 months
  Total rate of definite or probable stent thrombosis
Peri-Procedural Complications | 30 Days
  Rate of peri-procedural complications defined as angiographic complications in the study vessel.
Stroke | 30 Days
  Rate of disabling stroke
Bleeding | 30 Days
  Rate of Major bleeding
Kidney Injury | 30 Days
  Rate of Acute kidney injury (AKI)
Patient Reported Health Status - SAQ-7 | Baseline, Day 30 and 12 Months
  Seattle Angina Questionnaire (SAQ-7)
Patient Reported Quality of Life - EQ-5D | Baseline, Day 30 and 12 Months
  EuroQol Group EQ-5D-5L
Procedure Time | 24 hours
  Total time from arterial access to removal of last catheter in minutes
Contrast Dose | 24 hours
  Total amount of contrast used in ml
Radiation Dose | 24 hours
  Total amount of radiation in Gy
Resource utilization | 24 hours
  Hospital costs will be assessed for all patients based on procedural and index hospitalization resource utilization and standard US costs for each resource (including procedural time).
Cost-effectiveness | 12 Months
  Cumulative healthcare cost in dollars for every major adverse event avoided
FFRangio Usability | 24 hours
  Ability to conduct the FFRangio assessment without any system malfunction
Pressure Wire Usability | 24 hours
  Ability to conduct the pressure wire based assessment without any system malfunction

CONTACTS AND LOCATIONS:
Overall Officials: Ajay J Kirtane, MD, SM, Study Chair — NewYork-Presbyterian/Columbia University Irving Medical Center; William F Fearon, MD, Principal Investigator — Stanford University; Allen Jeremias, MD, MSc, Principal Investigator — St. Francis Hospital & Heart Center; Martin B Leon, MD, Study Chair — NewYork-Presbyterian/Columbia University Irving Medical Center
Locations (51):
- United States (43):
  - University of California San Diego Health, La Jolla, California
  - VA- Long Beach Healthcare, Long Beach, California
  - Keck Medicine of USC, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - VA - Palo Alto Healthcare, Palo Alto, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - St. Joesph's Medical Center, Stockton, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - HCA Florida JFK Hospital, Atlantis, Florida
  - Cardiac & Vascular Institute, Gainesville, Florida
  - HCA Florida Largo Hospital, Largo, Florida
  - HCA Florida Northside Hospital, St. Petersburg, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Archbold Hospital, Thomasville, Georgia
  - Carle Foundation Hospital, Urbana, Illinois
  - Ascension Via Christi St. Francis, Wichita, Kansas
  - Kansas Heart Hospital, Wichita, Kansas
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - TidalHealth, INC, Salisbury, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Ascension St. John Hospital, Detroit, Michigan
  - Metropolitan Heart Vascular Institute, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cardiac Associates Research, Tupelo, Mississippi
  - Mountainside Medical Center, Montclair, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - New York Presbyterian Methodist Hospital, Brooklyn, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center / New York Presbyterian Hospital, New York, New York
  - New York Presbyterian / Weill Cornell Medical Center, New York, New York
  - Northwell Health (Lenox Hill, North Shore, South Shore, Huntington, Staten Island)), New York, New York
  - St. Francis Hospital and Heart Center, Roslyn, New York
  - Ellis Hospital, Schenectady, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Mount Carmel Health System, Columbus, Ohio
  - Lehigh Valley Health, Allentown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas
  - HCA Methodist Healthcare of San Antonio, San Antonio, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
- Rabin Medical Centre, Petah Tikva, Israel
- Japan (4):
  - Gifu Heart Center, Gifu
  - Kobe University, Kobe
  - Mie University Hospital, Osaka
  - Sakakibara Heart Institute, Tokyo
- Switzerland (2):
  - Hopitaux Universitaires Geneve (HUG), Geneva
  - centre hospitalier universitaire vaudois (CHUV), Lausanne
- Imperial College Healthcare, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Redfors B, Madhavan MV, Kirtane AJ, Fearon WF, Yeh RW, Cohen DJ, Al-Lamee R, Jeremias A, Witberg G, Sharma RP, Popma A, Kaki A, Froimovich A, Leon MB. FFRangio-guided versus pressure wire-guided PCI: design and rationale of the multicentre, randomised ALL-RISE trial. EuroIntervention. 2025 Aug 18;21(16):961-969. doi: 10.4244/EIJ-D-25-00200. PMID 40828315